CLINICAL TRIAL: NCT03640273
Title: The Study of Efficacy and Adverse Effects of Prapchompoothaweep Remedy Crude Drug and Loratadine for Treatment in Allergic Rhinitis Patients (Clinical Trials Phase II)
Brief Title: Efficacy and Adverse Effects of Prapchompoothaweep Remedy and Loratadine for Treatment in AR Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supasuta Leangpanich, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Thammasat
Record Dates: First submitted 2018-07-09; First posted 2018-08-21 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Allergic Rhinitis; Adverse Drug Event; Quality of Life
Keywords: Loratadine; Prapchompoothaweep; Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Drug-Related Side Effects and Adverse Reactions | interventions — Loratadine

STUDY DESIGN:
Intervention Model Description: this study is a double blind randomized controlled trial study. the volunteers will be divided into 2 groups. One is received Prapchompoothaweep crude drug capsule at 1,000 mg 3 times a day before meals and the other is received Loratadine 10 mg per day before meals. it takes 6 weeks to complete the project for each volunteers.
  Before enrolling, volunteers will stop using any anti-histamine drug for 1 week (wash-out period). All volunteers will be followed up in the 3rd and 6th week to evaluate the efficacy and adverse effect after received drugs.
  The researcher will record characteristic data such as gender, age, BMI, vital signs and symptoms . The adverse effect will be monitored by hematology test e.g. liver function test, renal function test, lipid profile and blood sugar test.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prapchompoothaweep (Experimental): Group 1 will be received Prapchompoothaweep remedy 1,000 mg for 3 times before meals (for 6 weeks).
  Interventions: Drug: Prapchompoothaweep remedy
- Loratadine (Experimental): Group 2 will be received Loratadine 10 mg per day before meals (for 6 weeks)
  Interventions: Drug: Loratadine 10 Mg

INTERVENTIONS:
Drug: Prapchompoothaweep remedy — Take Prapchompoothaweep remedy capsule at 1,000 mg for 3 times a day before meals.
  Arms: Prapchompoothaweep
Drug: Loratadine 10 Mg — Take Loratadine 10 mg once a day before meals.
  Arms: Loratadine

SUMMARY:
1. To compare the effectiveness of Prapchompoothaweep crude drug at 3,000 mg per day and Loratadine 10 mg per day for treatment in Allergic Rhinitis patients. (Clinical Trial Phase II)
2. To evaluate the safety and adverse effect of Prapchompoothaweep crude drug at 3,000 mg and Loratadine 10 mg for Allergic Rhinitis patients.

DETAILED DESCRIPTION:
this study is a double blind randomized controlled trial study.

the volunteers will be divided into 2 groups. One is received Prapchompoothaweep crude drug capsule at 1,000 mg 3 times a day before meals and the other is received Loratadine 10 mg per day before meals. it takes 6 weeks to complete the project for each volunteers.

Before enrolling, volunteers will stop using any anti-histamine drug for 1 week (wash-out period). All volunteers will be followed up in the 3rd and 6th week to evaluate the efficacy and adverse effect after received drugs.

The researcher will record characteristic data such as gender, age, BMI, vital signs and symptoms . The adverse effect will be monitored by hematology test e.g. liver function test, renal function test, lipid profile and blood sugar test.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-70 years old.
* Patients with history of allergic rhinitis based on ARIA guidelines. (itching and nasal obstruction, watery nasal discharge, sneezing ,congestion)
* Patients with moderate allergic rhinitis was diagnosed by physicians.
* Have no nasal septum perforation, nasal polyp or sinus surgery.
* Have no serious medical conditions: Heart disease, Liver disease, Renal disease, Hypertension, Peptic Ulcer and Gastroesophageal reflux disease (GERD), severe Asthma, Tuberculosis.
* Have normal range of Hematology test for Liver and Renal function.
* No Pregnant or Lactation.
* Do not taking a medicine constantly.
* Volunteers are willing to participate this study.

Exclusion Criteria:

* Allergic reactions to Prapchompoothaweep remedy and Loratadine.
* Allergic reaction to dairy products.
* Have severe urticaria and anaphylaxis.
* Have a serious condition of immunodeficiency disease: HIV in the previous month before being recruited in the study.
* Participate in another study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-06-24 (Actual)

PRIMARY OUTCOMES:
Nasal cavity Change from baseline at 6 weeks | week-0, week-3 and week-6
  Using an Acoustic Rhinometry to evaluate nasal symptoms

SECONDARY OUTCOMES:
Assessment of well-being of volunteer that change from baseline at 6 weeks. | week-0, week-3 and week-6
  Using Rhinoconjunctivitis Questionnaire of Life (Thai Version copyright by Chaweewan Bunnag MD) This questionnaire is designed to find out how your health and well-being have been affected by rhinoconjunctivitis. score including 1-5 score; 1 = not at all, 2 = Slightly, 3 = moderately, 4 = A lot and 5 = Extremely.
Nasal symptoms Change from baseline at 6 weeks. | week-0, week-3 and week-6
  Using Total Nasal Symptom Score Questionnaire. This questionnaire is designed to estimate how severe of your nasal symptom. the questionnaire including the question of 4 symptom of Allergic Rhinitis; sneezing, nasal congestion, nasal itching and runny nose. the score was divided in 4 mark, 0-not at all, 1=slightly, 2=moderate,3=severe.
Renal Function Change from baseline at 6 weeks. | week-0, week-3 and week-6
  to evaluate the adverse events by hematology test of renal function which including BUN (mg/dL) and Creatinine (mg/dL). Normal range of BUN and Creatinine are 7.0-18.0 mg/dL and 0.67-1.17 mg/dL respectively.
Liver Function Change from baseline at 6 weeks. | week-0, week-3 and week-6
  to evaluate the adverse events by hematology test of liver function which including AST (U/L), ALT (U/L), Total Alkaline Phosphatase (U/L), total bilirubin (mg/dl), direct-bilirubin (mg/dl), Globulin (g/dl), Albumin (g/dl) and Total protein (g/dl).
  Normal range of AST, ALT, Alkaline Phosphatase, total bilirubin, direct-bilirubin, globulin, albumin and total protein are 16-37 U/L, 16-63 U/L, 46-116 U/L, 0.2-1.0 mg/dl, 0.0-0.2 mg/dl, 1.5-3.5 g/dl, 3.4-5.0 g/dl and 6.4-8.2 g/dl respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Effectiveness (Nasal Cavity, Nasal Score, Well-being) and Safety (Hematology test) of Prapchompoothaweep and Loratadine in Allergic Rhinitis patients.